CLINICAL TRIAL: NCT00492050
Title: Primary Treatment of Waldenstrom's Macroglobulinemia With Bortezomib (Velcade) and Rituximab (Rituxan) Followed by Autologous Stem Cell Collection
Brief Title: Bortezomib and Rituximab for Patients With Waldenstrom's Macroglobulinemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0733; NCI-2012-01498 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2022-05-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: Waldenstrom's Macroglobulinemia; Macroglobulinemic Lymphoma; Stem Cell Collection; Bortezomib; LDP-341; MLN341; PS-341; Velcade; Rituximab; Rituxan
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Bortezomib; Rituximab; Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bortezomib + Rituximab (Experimental): Bortezomib 1.6 mg/m^2 IV Weekly on Days 1, 8, 15 and 22. Rituximab 375 mg/m^2 IV on Day 8 and 22. Valacyclovir 500 mg orally daily (or acyclovir 200 mg orally twice daily).
  Interventions: Drug: Bortezomib; Drug: Rituximab; Drug: Valacyclovir

INTERVENTIONS:
Drug: Bortezomib — 1.6 mg/m^2 IV Weekly on Days 1, 8, 15 and 22.
  Other Names: Velcade; LDP-341; MLN341; PS-341
Drug: Rituximab — 375 mg/m^2 IV on Day 8 and 22.
  Other Names: Rituxan
Drug: Valacyclovir — 500 mg orally daily (or acyclovir 200 mg orally twice daily)
  Other Names: Valtrex

SUMMARY:
The main goal of this clinical research study is to learn if Velcade ® (bortezomib) given with rituximab can help to control WM. This drug combination will allow researchers to collect your stem cells in case it is possible to transplant the stem cells as treatment if your WM gets worse. Researchers will also look at the safety and tolerability of this drug combination followed by treatment with other drug combinations.

DETAILED DESCRIPTION:
Bortezomib is designed to block a protein that plays a role in cell function and growth, which may cause cancer cells to die.

Rituximab is designed to attach to cancer cells, which may cause them to die.

Cyclophosphamide, vincristine, doxorubicin, and cladribine are designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Dexamethasone is designed to decrease inflammation. It is also used to treat certain forms of cancer.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. The tests may be performed within 28 days of starting the study drug. You will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate), height, and weight. Your medical history will be recorded. You will be asked to fill out a questionnaire regarding any neuropathy (nerve problems) you may have. The questionnaire will take about 1 minute to complete. You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). You will also have blood (about 4-5 teaspoons) drawn one time and urine collected (over 24 hours) to check the status of your WM. This blood is also used to screen for hepatitis. You will have an x-ray of your chest. You will have computed tomography (CT) scans of your abdomen and pelvis to see which part of your body is involved with WM. If your chest x-ray is positive, you will also have a CT scan of your chest. Women who are able to have children must have a negative blood (about 2 teaspoons) or urine pregnancy test before starting the study. You will also have a bone marrow aspiration and biopsy. To collect a bone marrow aspirate/biopsy, an area of the hip bone will be made numb with an anesthetic, and a small amount of bone marrow and bone will be withdrawn through a large needle.

If you are found to be eligible to participate in this study, you will begin taking the study drugs. You will be given two 35-day cycles of bortezomib and rituximab. Bortezomib will be given through a needle in a vein over 3-5 seconds on Days 1, 8, 15, and 22. Rituximab will also be given through a vein on Days 8 and 22. The first rituximab infusion (by vein) usually takes 6-8 hours. Later infusions are generally shorter, taking about 4 hours to complete. While you are receiving bortezomib/rituximab (for 2-3 months), valacyclovir (an anti-viral drug) is taken by mouth, once a day.

During the study, before each dose of bortezomib, you will have blood (about 2 teaspoons each time) drawn for routine tests. Your vital signs will be measured. You will be asked about any side effects you may have experienced. You will also be asked to answer the questionnaire about any neuropathy you may have.

Stem cells are the cells from which all blood cells develop. If you respond to the first 2 cycles of bortezomib/rituximab, you will then have some of your stems cells collected. You will have to sign a separate consent form that describes this procedure and its risks. After the stem cell collection, 1 cycle of cladribine, cyclophosphamide, and rituximab will be given. Cladribine will be given through a vein once a day over 2 hours on Days 1-5. Cyclophosphamide is taken by mouth, twice a day on Days 1-5, and rituximab is given through a vein once a week for 4 weeks.

If you do not respond to the first cycle of bortezomib/rituximab, you will be taken off the study.

If you respond to the first but do not respond to the second cycle of bortezomib/rituximab, you will receive a third cycle. The bortezomib/rituximab will be given in the same manner as your first 2 cycles.

If you respond to the third cycle of bortezomib/rituximab, you will have some of your stems cells collected. After the stem cell collection, 1 cycle of cladribine, cyclophosphamide, and rituximab will be given. Cladribine will be given through a vein once a day over 2 hours on Days 1-5. Cyclophosphamide is taken by mouth, twice a day on Days 1-5, and rituximab is given through a vein once a week for 4 weeks.

If you do not respond to the third cycle of bortezomib/rituximab, you will be given a chemotherapy regimen containing the drugs rituximab, cyclophosphamide, vincristine, and doxorubicin, together with dexamethasone. This combination is known as modified R-Hyper-CVAD. Rituximab will be given through a vein over about 4 hours on Day 1 only. Cyclophosphamide will be given through a vein every 12 hours on Days 1-4. Doxorubicin and vincristine will be given through a vein continuously over 24 hours on Days 1-4. Dexamethasone is taken by mouth daily on Days 1-4, 9-12, and 17-20.

If a partial response is seen with modified R-Hyper-CVAD, you will have some of your stem cells collected. You will receive 1 cycle of cladribine, cyclophosphamide, and rituximab. Cladribine will be given through a vein once a day over 2 hours on Days 1-5. Cyclophosphamide is taken by mouth, twice a day on Days 1-5, and rituximab is given through a vein once a week for 4 weeks.

About 1 week before the start of each cycle of chemotherapy, you will have blood (about 4-5 teaspoons) drawn for routine tests and to see how your WM is responding. You may also need to collect your urine over 24 hours, depending on if the first test was initially positive or not. You will also have a complete physical exam, including measurement of vital signs, height, and weight.

If your CT scans were positive initially, you will need to have them repeated after 2 cycles of bortezomib/rituximab and then every 6 months. Once you have a partial response confirmed by CT scans, you will not need to repeat the CT scans anymore.

If your disease does not respond to modified R-Hyper-CVAD, you will be taken off the study.

Responding participants will be followed at least every 6 months for the first 36 months (from the end of therapy). After that, you will be followed at least once a year unless the disease gets worse and needs to be re-treated. For the follow-up evaluations, you will have a physical exam, including measurement of vital signs. Blood (about 4 tablespoons) will be drawn for routine tests. Blood (about 4-5 teaspoons) and urine (over 24 hours) will be collected to check the status of your WM. If the x-rays and/or CT scans done at the beginning of the study were positive, you will have repeat x-rays and/or CT scans.

For patients who have not had a partial response, follow-up evaluations will be at least every 3 months. You will have a physical exam, including measurement of vital signs. Blood (about 4 tablespoons) will be drawn for routine tests. Blood (about 4-5 tablespoons) and urine (over 24 hours) will be collected to check the status of your WM.

You will be taken off the study if you do not have a partial or complete response following 3 cycles of bortezomib/rituximab and 2 cycles of modified R-Hyper-CVAD. You will be taken off the study if the disease gets worse after all planned therapy that the study doctor feels requires repetition. You will be taken off the study if intolerable side effects occur. You will be taken off the study if treatment with bortezomib is delayed for more than 2 weeks. You will be taken off the study if you develop certain other illnesses, or if there are certain changes in your health that the study doctor decides may make further treatment with the study drugs to be unacceptable.

Once you are taken off the study, you will have an end-of-study visit. At this visit, a physical exam, including measurement of vital signs, height, and weight will be performed. You will be asked about any side effects that you may have experienced. You will be asked to answer the questionnaire regarding any neuropathy you may have. Blood (about 4-6 teaspoons) will be drawn for routine tests and to check the status of your WM. You will need to collect your urine over 24 hours to see how your WM is responding. If your initial CT scans showed lesions that appear to be caused by WM, you will have a CT scan repeated at this time.

If you have had a partial or complete response at the end of all planned therapy, you will need to return to the clinic for follow-up visits at least once every 6 months for the first 36 months (from the end of therapy). After that, you will have follow-up visits at least once a year, unless the disease gets worse and re-treatment is necessary. At the follow-up visits, you will have a physical exam, including measurement of vital signs, height, and weight. You will be asked about any side effects that you may have experienced. Blood (about 4-6 teaspoons) will be drawn for routine tests and to check the status of your WM. Depending on the results of your original urine tests, you may need to collect your urine over 24 hours to see how your WM is responding. If your initial CT scans showed lesions that appear to be caused by WM, you will have CT scans and an x-ray of your chest repeated at this time.

This is an investigational study. Cyclophosphamide, vincristine, doxorubicin, and rituximab are commercially available and FDA-approved for treatment of Waldenstrom's macroglobulinemia. Bortezomib, dexamethasone, cladribine, and the drug combinations used in this study have been authorized for use in research only. Bortezomib has been FDA approved and it is registered in Europe for the treatment of multiple myeloma patients who have received at least one prior therapy. Tests/procedures that are required for this study are considered to be part of your routine medical care. Up to 38 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic macroglobulinemic lymphoma who have had no prior treatment, or whose prior treatment has been limited to steroids and/or alpha-interferon, are eligible. Macroglobulinemic lymphoma includes patients with either biopsy proven clonal lymphocytic or lymphoplasmacytic proliferation and monoclonal IgM. Also included are symptomatic patients with clonal proliferation producing a pathologic monoclonal IgM that causes cryoglobulinemia, peripheral neuropathy or cold agglutinin hemolytic anemia.
2. Patients must have acceptable liver function (total bilirubin < 2.5mg/dL) and renal function (creatinine < 2.0mg/dL). Patients with impaired renal function will only be included if the renal failure is secondary to macroglobulinemic lymphoma (i.e. Bence Jones proteinuria, cryoglobulinemia, ureteral obstruction due to mass) that might reverse with improvement of disease.
3. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
4. Male subject agrees to use an acceptable method for contraception for the duration of the study.
5. Patients must voluntarily sign an informed consent form indicating that they are aware of the investigational nature of the study, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future care.
6. Patient has a heart rate (HR) of greater than or equal to 50 bpm.

Exclusion Criteria:

1. Patient has a platelet count of <30x10^9/L within 28 days before enrollment unless due to >/= 75% marrow infiltration by macroglobulinemic lymphoma or splenomegaly.
2. Patient has an absolute neutrophil count of <1.0x10^9/L within 28 days before enrollment unless due to >/= 75% marrow infiltration by macroglobulinemic lymphoma.
3. Patient has a calculated or measured creatinine >/= to 2.0mg/dL on baseline evaluation. Patients with impaired renal function will only be included if the renal failure is secondary to macroglobulinemic lymphoma (i.e. Bence Jones proteinuria, cryoglobulinemia, ureteral obstruction due to mass).
4. Patient has >/= Grade 2 peripheral neuropathy on baseline evaluation.
5. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
6. Patient has hypersensitivity to boron, mannitol, or murine proteins.
7. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum or urine Beta -human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
8. Patient has received other investigational drugs within 14 days before enrollment
9. Patient has a serious medical or psychiatric illness that is likely to interfere with participation in this clinical study.
10. Eastern Cooperative Oncology Group (ECOG) performance status of > 2.
11. Patient with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled. Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for > 5 years and are considered by their physician to be at less than 30 % risk of relapse.
12. Patient with a lifetime cumulative dose of > 450 mg/m^2 of anthracyclines.
13. Patients with an active hepatitis B infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-08-02 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2026-06-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sheeba Thomas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 2006- March 2013
Pre-assignment Details: 46 Participants consented, 9 screen failures.
Period: Overall Study
Arm/Group | Bortezomib + Rituximab
Started ((Additonal cycle 3); Bortezomib 1.6 mg/m2, Rituximab 375 mg/m2 (1 additional cycle)) | 37
Inadequate Response to First Two Cycles | 25
Inadequate Response to First 3 Cycles (Rituximab 375 mg/m^2, Cyclophosphamide 100 mg/m^2, Doborubicine 9 mg/m^2/day, dexamethasone 40 mg/day (2 cycles)) | 12
If Adequate Response to First Two Cycles-participants Proceed to Stem Cell Collection (+ 1 cycle of 2CdA 3.0 mg/m2, cyclophosphamide 60 mg/m2, rituximab 375 mg/m2) | 30
Completed | 28
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 3
Not completed — Unable to collect SCT | 2
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Bortezomib 1.6 mg/m^2 IV Weekly on Days 1, 8, 15 and 22. Rituximab 375 mg/m^2 IV on Day 8 and 22. Valacyclovir 500 mg orally daily (or acyclovir 200 mg orally twice daily).
  Bortezomib: 1.6 mg/m^2 IV Weekly on Days 1, 8, 15 and 22.
  Rituximab: 375 mg/m^2 IV on Day 8 and 22.
  Valacyclovir: 500 mg orally daily (or acyclovir 200 mg orally twice daily)
Arm/Group | All Participants
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 61 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 37
Newly diagnosed patient with Waldenstrom Macroglobulinemia with no prior treatment [Count of Participants; unit: Participants] | 37

OUTCOME MEASURES:

1. Primary Outcome: Response Rate After 2 Cycles of Treatment With Bortezomib and Rituximab
Description: Partial response (PR) defined as at least > 50 % reduction of serum monoclonal IgM concentration determined by protein electrophoresis, > 50% decrease in adenopathy / organomegaly on physical examination or on CT scan, and no new symptoms or signs of active disease. Complete response (CR) defined as a disappearance of serum and urine monoclonal protein determined by immunofixation, absence of malignant cells in bone marrow determined by histologic evaluation, resolution of adenopathy/organomegaly (confirmed by computed tomography [CT] scan), and no signs or symptoms attributable to WM. Stable disease defined as neither grown nor shrunk; the amount of disease has not changed.Participants will be followed for < 6 months after receiving bortezomib/rituximab or rituximab-modified hyper-CVAD to be considered unresponsive to therapy in accordance with the guidelines of the Consensus Panel of the Third International Workshop on Waldenstrom's Macroglobulinemia.
Time Frame: After 2 (35 day) cycles of treatment
Population: 1 subject didn't complete 2 cycles of therapy and isn't evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 36
Participants
  Stable Disease | 20
  Partial Response | 11
  Progressive Disease | 2
  No Response | 3

2. Primary Outcome: Response Rate After 3 Cycles of Treatment With Bortezomib and Rituximab
Description: Partial response (PR) defined as at least > 50 % reduction of serum monoclonal IgM concentration determined by protein electrophoresis, > 50% decrease in adenopathy / organomegaly on physical examination or on CT scan, and no new symptoms or signs of active disease. Complete response (CR) defined as a disappearance of serum and urine monoclonal protein determined by immunofixation, absence of malignant cells in bone marrow determined by histologic evaluation, resolution of adenopathy/organomegaly (confirmed by computed tomography [CT] scan), and no signs or symptoms attributable to WM. Stable disease defined as neither grown nor shrunk; the amount of disease has not changed. Participants will be followed for < 6 months after receiving bortezomib/rituximab or rituximab-modified hyper-CVAD to be considered unresponsive to therapy in accordance with the guidelines of the Consensus Panel of the Third International Workshop on Waldenstrom's Macroglobulinemia.
Time Frame: After 3 (35 day) cycles of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 25
Participants
  Stable Disease | 7
  Partial Response | 16
  No Response | 2

3. Primary Outcome: Participants Ability to Collect Stem Cells After Treatment With Bortezomib and Rituximab
Description: Number of Participants who were able to collect stem cells successfully or unable to collect after treatment with bortezomib and rituximab.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 37
Participants
  Participants Collected Successfully | 30
  Participants Unable to Collect | 7

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dosage up to 5 years
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 14/37
Other Adverse Events (participants affected / at risk) | 14/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=37)
Anemia (Blood and lymphatic system disorders) | 2
Hypotension (Cardiac disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Elevated Alkaline Phosphate (Gastrointestinal disorders) | 1
Fever (Infections and infestations) | 1
Gram negative bacteremia (Infections and infestations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Neutrophenic fever (Infections and infestations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 1
Spetic shock (Infections and infestations) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Visual changes (General disorders) | 1
Hyperviscosity (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=37)
Fatigue (General disorders) | 6
Diarrhea (Gastrointestinal disorders) | 3
Pain (joint) (Musculoskeletal and connective tissue disorders) | 4
Pain (muscle) (Musculoskeletal and connective tissue disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 4
Dizziness (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
BUN increase (Renal and urinary disorders) | 1
Creatinine increase (Renal and urinary disorders) | 1
Dry eye (Eye disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Peripheral Edema (Vascular disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neuopathy (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT00492050/Prot_SAP_000.pdf